CLINICAL TRIAL: NCT00849368
Title: Dose-effect Relationship Between Allopurinol, Azathioprine and 6-thioguanine Nucleotide Levels (6-TGN) in Inflammatory Bowel Disease Patients.
Brief Title: Azathioprine & Allopurinol in Inflammatory Bowel Disease Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Alexander Jetter, PD Dr. med., University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHA-08-AZA/ALLO-01
Record Dates: First submitted 2008-09-02; First posted 2009-02-23 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Azathioprine; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azathioprine / Allopurinol (Experimental): Single arm study: Dose escalations as described.
  Interventions: Drug: Azathioprine / Allopurinol

INTERVENTIONS:
Drug: Azathioprine / Allopurinol — Both drugs are applied orally. A pre-specified dose escalation regimen will be chosen.
  Azathioprine: Imurek (R) 50 mg and 25 mg tablets
  Allopurinol: Mephanol (R) 100 mg tablets
  Other Names: Azathioprine: Imurek (R) 50 mg and 25 mg tablets; Allopurinol: Mephanol (R) 100 mg tablets

SUMMARY:
Main Study Objectives:

The study is conducted to

* evaluate the minimal allopurinol and azathioprine doses that, in combination, produce therapeutic 6-TGN levels
* evaluate the safety and tolerability of the different allopurinol/azathioprine dose levels
* assess if concomitant allopurinol affects TPMT activity
* assess the clinical efficacy of concomitant allopurinol-azathioprine therapy in the included patients

ELIGIBILITY:
Inclusion criteria:

* Able and willing to give written informed consent before any trial-specific procedures are performed
* Signed informed consent form
* Age 18 to 65 years at study entry
* Body Mass Index 18 - 30 kg/m2
* Confirmed diagnosis of either CROHN's disease or ulcerative colitis prior to study enrollment by combinations of clinical, endoscopic and histologic criteria generally accepted for CD and UC
* Normal TPMT activity > 30 nmol MTG/gHb x h
* Insufficient disease control despite adequate therapy with corticosteroids and/or salicylic acid derivatives, and/or two or more episodes with steroid-requiring disease activity per year, and/or recurrence of disease activity at steroid doses below 15 mg prednisone equivalent, and/or recurrence within 6 weeks after steroid withdrawal.

Exclusion criteria:

* Subjects with confirmed or suspected hypersensitivity towards the study medication
* Contemporaneous participation in any other study
* Females only: pregnancy
* Females only: breast-feeding
* Prior thiopurine therapy
* Current and previous immunosuppressive therapy except corticosteroids (e.g. methotrexate, cyclosporine, mycophenolate mofetil, tacrolimus, infliximab or other TNF-alpha blocker therapy) within 3 months before the first drug intake
* Subjects with any clinically relevant comorbidity beyond the diagnosis of CROHN's disease or ulcerative colitis (as based on extensive medical history, physical examination, vital signs, routine laboratory screen and 12-lead ECG)
* Haemoglobin < 12 g/dl at the screening examination
* Leucocytes < 3 x 10E3/µl at the screening examination
* Lymphocytes < 1.5 x 10E3/µl at the screening examination
* Thrombocytes < 140 x 10E3/µl at the screening examination
* Renal disease (creatinine clearance < 60 ml/min, assessed with MDRD formula), history of serious renal disease
* Liver disease (GGT, alkaline phosphatase, ALAT, ASAT > 2 times the upper limit of normal reference, known or suspected liver cirrhosis)
* Known or suspected malignancies of any kind
* Known or suspected active infections, serious infections in the preceding 3 months
* Active, acute or chronic, or history of, prior hepatitis B infection confirmed by a positive hepatitis B serology (positive HBsAg, Anti-HBc). Patients with a positive hepatitis C screening test (positive anti-HCV). Patients with a positive HIV testing (positive HIV 1 / 2 antibody tests)
* Active varicella zoster infection (chickenpox, shingles)
* Known or suspected symptomatic bowel stenoses or strictures, and patients who had a small bowel resection
* Subjects who are known or suspected not to be capable of understanding and evaluating the information that is given to them as part of the formal information policy (informed consent), in particular regarding the risks and discomfort to which they will be exposed
* Subjects who are known or suspected not to comply with the study directives and / or known or suspected not to be reliable or trustworthy
* Subjects who are not willing to comply with the instructions and duties concerning the subject insurance
* Women of childbearing age and potential who are not willing or capable to use acceptable methods of contraception (oral contraceptives, condoms, diaphragms, intrauterine devices) during the entire study and for up to three months after the end-of-study evaluation.
* Male patients who do not use acceptable barrier methods of contraception (condoms) during the entire course of the study and up to three months after the end-of-study evaluation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Quantification of trough concentrations of 6-TGN and 6-MMPN in erythrocytes using HPLC at each dose level. | three times per cycle

SECONDARY OUTCOMES:
Dose escalation: Assessment of the percentage of patients who are in the desired therapeutic range on day 23-25 and on day 26-28 of each dose level. | once per cycle
Efficacy: Change in disease activity score in relationship to the dose level attained. | once per cycle
TPMT activity assessment | once per cycle
Safety and Tolerability: Medical history, adverse events and well-being; laboratory screen, physical examination, vital functions: blood pressure, heart rate, body temperature | screening, up to three times per cycle, follow-up

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Alexander Jetter, MD, Principal Investigator — Division of Clinical Pharmacology and Toxicology, University Hospital Zürich, 8091 Zürich, Switzerland
Locations (1):
- Division of Clinical Pharmacology and Toxicology, University Hospital Zurich, Zurich, Switzerland